CLINICAL TRIAL: NCT05688774
Title: Study of Progression of Hospitalized Community Acquired Pneumonia - Genetic Resistance and Susceptibility for the Evolution of Severe Sepsis in Patients With More Severe Preexisting Diseases and Immunosuppression to Complement the PROGRESS CAP Cohort
Brief Title: Study of Progression of Community Acquired Pneumonia in the Hospital in Patients With More Severe Preexisting Diseases and Immunosuppression
Acronym: PROGRESSCOMORB
Status: Recruiting | Type: Observational
Sponsor: Pneumonia Research Network on Genetic Resistance and Susceptibility for the Evolution of Severe Seps (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Leipzig (Other); Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROGRESS-COMORB
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pneumonia; Sepsis; Shock, Septic
Keywords: community ascquired pneumonia; CAP; disease progression
MeSH Terms: conditions — Pneumonia; Sepsis; Shock, Septic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from EDTA whole blood, RNA from stabilized whole blood, serum, citrate plasma, stabilized EDTA plasma, urin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumonia is a common infectious disease of the lung, often requiring treatment in the hospital. Clinical scoring systems are available, identifying patients not requiring hospitalization. However, the course of disease of patients in the hospital remains hard to predict. While most patients will recover quickly, some will, despite appropriate treatment, develop a severe course leading to sepsis and systemic responses resulting in organ dysfunction. The PROGRESS consortium aims to identify clinical, genetic, and other molecular markers and combinations there of predicting a severe course of pneumonia in the hospital. Such predictors will, for instance, support decisions on earlier transfer of patients to intensive care and thus improving outcome. PROGRESS-COMORB aims to extend findings from the previous PROGRESS study to patients with more severe preexisting conditions and immunosuppression.

DETAILED DESCRIPTION:
Pneumonia is a common infectious disease of the lung, often requiring treatment in the hospital. Clinical scoring systems are available, identifying patients not requiring hospitalization. However, the course of disease of patients in the hospital remains hard to predict. While most patients recover quickly, others will, despite appropriate treatment, develop a severe course leading to sepsis and systemic responses resulting in organ dysfunction. The PROGRESS consortium aims to identify clinical, genetic and other molecular markers and combinations there of predicting a severe course of pneumonia in the hospital. Such predictors will, for instance, support decisions on earlier transfer of patients to intensive care and thus improving outcome. PROGRESS-COMORB aims to extend findings from the previous PROGRESS study to patients with more severe preexisting conditions and immunosuppression.

In this observational, longitudinal case-cohort study, patients are enrolled within 48 hours of hospitalization (within 7 days for patients directly admitted to intensive care) and patient's progress is followed in much detail for up to six days thereafter. Further data are collected until discharge from the hospital. Patients are followed up on at days 28, 180, and 360 after enrollment.

Baseline assessment comprises sociodemographic, anamnestic, family history, and life-style information. Upon enrollment, Pneumonia Severity Index (PSI) and CURB-65 are determined. For the day of enrollment, up to six subsequent study days routine laboratory and clinical observations and information on therapy are documented as well as data for determining the Sequential Organ Failure Assessment (SOFA) score, Systemic Inflammatory Response Syndrome (SIRS) status, and organ dysfunction. Starting with enrollment, up to four consecutive sets of biomaterials are collected comprising serum, plasma, and materials for extraction of RNA. Blood for extraction of DNA is collected once.

Follow up comprises vital status, housing situation, recurrence of pneumonia, stroke, myocardial infarction, occurrence of diabetes and a quality of life questionnaire.

In the PROGRESS consortium, the transition (progression) from uncomplicated community-acquired pneumonia acquired pneumonia (uCAP) to severe CAP (sCAP) to CAP with severe sepsis or septic shock or multiple organ failure (ssCAP) is investigated. Previous work of the PROGRESS consortium led to the successful identification of an operationalization for the severity of CAP and causal pathomechanistic correlations, a clinical prognosis score, the assignment of altered molecules to dysfunctions of the respiratory tract, kidneys, coagulation, cardiovascular system, and liver, and a gene expression signature for early detection of patients at risk of developing ssCAP.

For the translation of findings from the PROGRESS-CAP study into clinical applicability, their applicability to CAP patients with immunosuppression or with more severe preexisting conditions has to be confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization with community acquired pneumonia (CAP) confirmed by pulmonary infiltrate in chest imaging
2. Valid informed consent form
3. Working diagnosis of CAP by enrolling physician
4. No hospitalization for any reason within 28 days prior to hospitalization for the current episode of CAP
5. At least 2 out of the five following clinical symptoms:

   * Fever
   * Cough
   * Purulent sputum
   * Shortness of breath or need for respiratory support
   * Crackling or rales on auscultation, dullness to percussion, or bronchial breathing
6. At least 1 of the following criteria

   * Known HIV infection or AIDS
   * Anti-tumor treatment within the past six months
   * Therapy with corticosteroids ≥ 20mg for ≥ 14 days before enrollment
   * Non-steroidal immunosuppressive therapy within the past six months
   * Cytostatic therapy within the past six months
   * Radiation therapy within the past six months
   * Bone marrow transplant received
   * Respiratory support at home via tracheostoma
   * Cystic fibrosis
   * Heart failure: New York Heart Association (NYHA) Stadium IV or HFrEF (defined as left ventricular ejection fraction <40%).
   * Decompensated liver disease (Child-Pugh class C)
   * Diabetes mellitus with HbA1c ≥ 8,5 %
   * End-stage renal disease requiring dialysis
   * Pulmonary hypertension (all classes) with mPAP > 20 mmHg (right heart catheter)

Exclusion Criteria:

1. Participation in this study at an earlier time
2. More than 48 hours in the hospital before enrollment (for patients directly to intensive care: more than 7 days)
3. Pregnancy
4. Breastfeeding
5. Active tuberculosis
6. Acute lung injury or acute respiratory distress syndrome for extrapulmonary reasons
7. Massive aspiration
8. Sepsis with extrapulmonary focus
9. Acute pulmonary embolism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized for treatment of community acquired pneumonia. Patients can be enrolled in general care, intensive care, and in emergency departments.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Worst measure of disease severity | Between enrollment and day six
  Disease severity is operationalized by the Sequential Organ Failure Assessment (SOFA-score).

SECONDARY OUTCOMES:
All cause mortality | up to one year after enrollment
disease-specific mortality | up to one year after enrollment
duration of hospitalization | up to one year after enrollment
duration of intensive care treatment | up to one year after enrollment
duration of ventilator assisted breathing | up to one year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Suttorp, MD, Principal Investigator — Charité Univerity, Berlin, Germany
Locations (10):
- Germany (10):
  - Charité - Universitätsmedizin Berlin, Medizinische Klinik m. S. Infektiologie und Pneumologie, Berlin
  - Humboldt-Klinikum Vivantes, Kardiologie und kons. Intensivmedizin, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Kardio-Pneumologie, Berlin
  - Städtisches Klinikum Dessau, Innere Medizin, Dessau
  - Universitätsklinikum Hamburg Eppendorf, Onkologisches Zentrum, Pneumologische Studienzentrale, Hamburg
  - Universitätsklinikum Leipzig, Klinik für Onkologie, Gastroenterologie, Hepatologie, Pneumologie, Leipzig
  - Klinikum St. Georg gGmbH, Klinik für Infektions-/Tropenmedizin und Nephrologie, Leipzig
  - Universitätsklinikum Gießen und Marburg, Klinik für Pneumologie und Anästhesie, Marburg
  - Universitätsklinikum Münster, Kardiologie 1, Münster
  - Diakoniekrankenhaus Rotenburg(Wümme)gGmbH, Zentrum für Pneumologie, Rotenburg (Wümme)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be made available after conclusion of the study. Participants can apply for clinical and molecular study data by sending structured project proposals to the PROGRESS board. The PROGRESS board will evaluate proposals for scientific quality, adherence to the limits set by patient's informed consent statements and by intellectual property regulations of the funding agency. Proposals shall not be denied without concrete reason.